CLINICAL TRIAL: NCT00596024
Title: Lutein and Oxidative Stress in Alzheimer's Disease - A Pilot Study
Brief Title: Lutein and Alzheimer's Disease Study
Acronym: LAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon Partnership for Alzheimer's Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAD; Alzheimer research fund
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Daily Lutein/zeaxanthin supplementation with a meal
  Interventions: Dietary Supplement: lutein/zeaxanthin
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: lutein/zeaxanthin — daily supplementation of lutein and zeaxanthin at dose of 12 mg/day
  Arms: 1
Dietary Supplement: placebo — placebo capsules with the same size and coating as those of lutein/zeaxanthin supplements without active ingredients
  Arms: 2

SUMMARY:
Oxidative damage by free radicals may be involved in causing Alzheimer's disease (AD). Free radicals may lead to death of nerve cells and decline in brain function. Certain antioxidants may suppress this free radical damage associated with AD. Carotenoids are a family of naturally occurring antioxidants that have important functions for human health. Carotenoids are known to reduce oxidative damage, but their effects have not been studied in AD patients.

The objective of the study is to examine whether lutein supplementation helps to reduce oxidative damage from free radicals in AD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderately severe Alzheimer's disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
oxidative damage markers | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States